CLINICAL TRIAL: NCT05095311
Title: The Effect of Cetirizine HCl on Exercise-induced Arterial Hypoxemia in Highly-trained Swimmers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The recruited population was no longer made available to participate in the study.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Robert Chapman, Principal Investigator, Indiana University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10766
Record Dates: First submitted 2021-06-19; First posted 2021-10-27 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Exercise-induced Arterial Hypoxemia
MeSH Terms: interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental group (Experimental): This subset of 12 individuals will complete all experimental study visits, and will ingest either 1) a placebo pill and placebo inhaler contents or 2) a cetirizine HCl pill (10 mg) and placebo inhaler contents in a randomized order and double-blind fashion.
  Interventions: Drug: Cetirizine HCl; Other: Placebo
- Selection pool (No Intervention): Twenty-four total individuals will be recruited for the initial portion of the study, and the aforementioned 12 (6 men, 6 women) will be a subset of the initial 24. The other 12 participants will not take part in further study.

INTERVENTIONS:
Drug: Cetirizine HCl — Eight participants will be administered 10 mg of cetirizine HCl to examine whether this drug can improve their oxyhemoglobin saturation during exercise.
  Other Names: Zyrtec
  Arms: Experimental group
Other: Placebo — The placebo pill is a sugar-free gelatin pill casing. The placebo inhaler contains isotonic saline.
  Arms: Experimental group

SUMMARY:
Exercise-induced arterial hypoxemia (EIAH), a reduced amount of oxygen in the arterial blood during exercise, has been observed in otherwise healthy, highly-trained endurance athletes during exercise at sea level. The extent of the arterial deoxygenation may be influenced by a histamine-mediated inflammatory response at the pulmonary capillary-alveolar membrane limiting oxygen diffusion. Moreover, while EIAH has been routinely explored in running and cycling, swimming is understudied despite potential mechanistic avenues which may put swimmers at further risk for EIAH. The purpose of this study is threefold: 1) to determine whether highly-trained swimmers experience EIAH during submaximal and maximal exercise, 2) to determine the extent to which histamine release influences oxyhemoglobin saturation during swimming exercise, and 3) to determine whether cetirizine HCl (CH), an H1-receptor competitive inhibitor, can improve oxyhemoglobin saturation during submaximal and maximal swimming exercise. Twenty-four (12 men, 12 women) highly-trained swimmers will complete an intense swimming protocol to assess the histamine response to intense exercise. A subset with the highest histamine responses will participate in three additional sessions (placebo, NS, and CH conditions) which will include a swimming aerobic capacity test and 5-minutes of swimming at both 70 and 85% of their maximal oxygen uptake.

DETAILED DESCRIPTION:
For the first testing session, participants will report to the Indiana University Human Performance Laboratory to complete a medical screening and, if willing, consent to the procedures of the study. The medical screening will include measurements of height, weight, resting heart rate, resting blood pressure, and resting pulmonary function along with a health history questionnaire.

The second testing session consists of an assessment of risk factors for development of EIAH, specifically changes in blood biomarkers pre- and post-swimming exercise. Participants will report to the Counsilman-Billingsley Aquatics Center and complete an exercise protocol designed to elicit an inflammatory response. Venous blood draws will be performed to assess participants' pre-exercise complete blood count and pre- and post-intense exercise concentrations of plasma IL-1β, IL-8, plasma histamine, whole blood histamine, and histamine release. Measurements of hemoglobin concentration and hematocrit will also be performed pre- and post-exercise in order to correct biomarker concentrations for fluid loss during exercise. Swimmers of each sex that exhibit the largest histamine release will be selected for further study until at least four swimmers of each sex complete all three experimental trials.

Twelve swimmers (n = 6 men, n = 6 women) will be selected for further trials. Those selected for further study will visit the Human Performance Laboratory on two occasions separated by at least 48 hours and no more than 60 days. Apart from receiving a placebo (PL) or drug treatment (cetirizine HCl, CH) prior to exercise, participants will perform identical protocols on each visit to the laboratory. Participants will report to the lab and consume either a placebo or CH pill, followed by a health history update questionnaire and their resting pulmonary function will be measured. Participants will then complete a self-selected warm-up that will be standardized across all testing sessions, followed by instrumentation. The exercise protocol beings with a progressive swimming test to maximum aerobic capacity (V̇O2max) in a swimming flume, followed by two constant load work bouts at approximately 70 and 85% of the previously recorded HRmax while peripheral capillary oxyhemoglobin saturation (SpO2) is continuously monitored. Participants will receive a 20-min break between each work bout. Drug treatments will be assigned in a double-blind, randomized crossover fashion such that each participant receives each treatment. Concentrations of plasma histamine, whole blood histamine, and histamine release will be assessed from pre- and post-exercise blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-35 years old
* Current collegiate or professional swimmer
* Currently training at least 300 minutes per week
* Self-reported to be healthy

Exclusion Criteria:

* Not within defined age range
* Current diagnosis of or using medication for:

  * Severe allergies
  * Asthma
  * Exercise-induced asthma
  * Exercise-induced bronchoconstriction
* Pulmonary function test considered to be abnormal (defined as forced vital capacity (FVC) <80% of predicted, forced expiratory volume in one second (FEV1) <80% predicted, and/or FEV1/FVC ratio >5% of the predicted ratio)
* Hypertension during screening (systolic blood pressure >139 or diastolic blood pressure >89)
* Current tobacco or electronic cigarette use or consistent use within the last 2 years
* A contraindication for use of nedocromil sodium:

  * Previous adverse reaction to nedocromil sodium or a similar medication
  * Use of fast-acting, inhaled insulin
* A contraindication for use of cetirizine HCl:

  * Previous adverse reaction to cetirizine HCl or a similar medication
  * Allergy to the food additives E218 or E216
  * An intolerance to or inability to absorb some sugars, such as lactose or sorbitol
  * Liver or kidney failure
  * Epilepsy or similar condition
  * A condition that makes urinating difficult
  * Use of midodrine or ritonavir
* Are pregnant or could possibly be pregnant by self-report
* Subjects with current, irregular menstrual cycles (amenorrhea) or who had irregular menstruation patterns for greater than one year
* People who answer 'yes' to any of the pre-participation screening questions on page one of the PAR-Q+ questionnaire.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Chapman, PhD, Principal Investigator — Professor
Locations (1):
- 1025 E Seventh St, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be published in the form of a dissertation document.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available upon degree certification (anticipated May 2022) and will be available indefinitely.
Access Criteria: The dissertation document will be publicly available.

REFERENCES:
- [Result] Coyle MA, Goss CS, Manz WJ, Greenshields JT, Chapman RF, Stager JM. Nedocromil sodium and diphenhydramine HCl ameliorate exercise-induced arterial hypoxemia in highly trained athletes. Physiol Rep. 2022 Jan;10(1):e15149. doi: 10.14814/phy2.15149. PMID 35001564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period lasted from March 2021 through April 2022. Participants were connected to the investigators through their coach, and participants were asked to schedule a screening visit (Visit 1) if desired.
Pre-assignment Details: The experimental arm of the study was limited to those participants who wanted to continue with the study and responded to correspondence from investigators.
Groups:
- Initial Phase Only: Twenty-four total individuals will be recruited for the initial portion of the study, and the aforementioned 12 (6 men, 6 women) will be a subset of the initial 24. The other 12 participants will not take part in further study.
- Initial Phase, Then Cetirizine HCl First, Then Placebo: This subset of 12 individuals will complete all experimental study visits, and will ingest either 1) a cetirizine HCl pill (10 mg) then 2) a placebo pill in double-blind fashion.
  Cetirizine HCl: Eight participants will be administered 10 mg of cetirizine HCl to examine whether this drug can improve their oxyhemoglobin saturation during exercise.
  Placebo: The placebo pill is a sugar-free gelatin pill casing.
- Initial Phase, Then Placebo First, Then Cetirizine HCl: This subset of 12 individuals will complete all experimental study visits, and will ingest either 1) a placebo pill then 2) a cetirizine HCl pill (10 mg) in double-blind fashion.
  Cetirizine HCl: Eight participants will be administered 10 mg of cetirizine HCl to examine whether this drug can improve their oxyhemoglobin saturation during exercise.
  Placebo: The placebo pill is a sugar-free gelatin pill casing.
Period: Overall Study
Arm/Group | Initial Phase Only | Initial Phase, Then Cetirizine HCl First, Then Placebo | Initial Phase, Then Placebo First, Then Cetirizine HCl
Started | 12 | 2 | 2
Completed | 5 | 2 | 2
Not Completed | 7 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Selection Pool | Total
Number analyzed (Participants) | 4 | 12 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 12 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (1.8) | 20.1 (1.9) | 20.1 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 12 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 12 | 16
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: liters] | 6.76 (0.91) | 6.87 (1.17) | 6.85 (1.09)
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] | 4.92 (0.67) | 5.40 (0.86) | 5.28 (0.82)
Forced Mid-Expiratory Flow (FEF25-75%) [Mean (Standard Deviation); unit: liters] | 3.88 (0.60) | 5.08 (1.11) | 4.78 (1.12)
Peak Expiratory Flow (PEF) [Mean (Standard Deviation); unit: liters per second] | 10.14 (1.75) | 9.21 (1.29) | 9.45 (1.42)

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Capillary Oxyhemoglobin Saturation
Description: SpO2 percentage measured via a standard bedside pulse oximetry unit
Time Frame: In the final minute of the aerobic capacity test and each of the two (70% and 85% of max) constant load trials in Visits 3 and 4 of the study
Population: These individuals are from the Experimental group.
Measure: Mean (Standard Deviation); unit: percent hemoglobin saturation
Groups:
- Cetirizine HCl: 10 mg of cetirizine HCl to examine whether this drug can improve their oxyhemoglobin saturation during exercise.
Arm/Group | Placebo | Cetirizine HCl
Number analyzed (Participants) | 4 | 4
percent hemoglobin saturation
  Aerobic capacity test | 96.8 (1.3) | 98.0 (1.8)
  70% constant load | 98.2 (1.8) | 98.5 (1.1)
  85% constant load | 98.8 (1.3) | 97.9 (1.4)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: There were no adverse events.
Groups:
- Initial Phase: Twenty-four total individuals will be recruited for the initial portion of the study, and the aforementioned 12 (6 men, 6 women) will be a subset of the initial 24. The other 12 participants will not take part in further study.
- Cetirizine HCl: This subset of 12 individuals will complete all experimental study visits, and will ingest either 1) a cetirizine HCl pill (10 mg) then 2) a placebo pill in double-blind fashion.
  Cetirizine HCl: Eight participants will be administered 10 mg of cetirizine HCl to examine whether this drug can improve their oxyhemoglobin saturation during exercise.
  Placebo: The placebo pill is a sugar-free gelatin pill casing.
- Placebo: This subset of 12 individuals will complete all experimental study visits, and will ingest either 1) a placebo pill then 2) a cetirizine HCl pill (10 mg) in double-blind fashion.
  Cetirizine HCl: Eight participants will be administered 10 mg of cetirizine HCl to examine whether this drug can improve their oxyhemoglobin saturation during exercise.
  Placebo: The placebo pill is a sugar-free gelatin pill casing.
Arm/Group | Initial Phase | Cetirizine HCl | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/16 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT05095311/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT05095311/ICF_003.pdf